CLINICAL TRIAL: NCT04356781
Title: Do (IgG) Variations in Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIPD) and MMN Patients Following Initial Intravenous Immunoglobulin (IVIg) Treatment Correlate with Ultimate Dosing
Brief Title: Do IgG Level Variations in CIDP and MMN Patients Following Initial Intravenous IVIg Treatment Correlate with Ultimate Dosing
Acronym: digG
Status: Completed | Type: Observational
Sponsor: Walton Centre NHS Foundation Trust (Other)
Collaborators: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: RG280-19
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Multifocal Motor Neuropathy (MMN); Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Keywords: CIDP, IgG, Immunoglobulin, IVIg, transfusion reaction
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Transfusion Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
CIDP and MMN are part of a group of chronic inflammatory conditions that affect the peripheral nervous system. In CIDP, there is chronic inflammation of the peripheral nerves and nerve roots leading to demyelination. The myelin sheath is vital in the rapid propagation of nerve impulses between the central nervous system and the peripheral sensory receptors and muscles. By definition CIDP must progress over 8 or more weeks and can either have a slowly progressive disease course or a relapsing course with periods of improvement. Patients typically present with a non-length dependent neuropathy that affects motor (i.e. weakness of proximal or distal muscles, fatigue, swallowing difficulty, double vision, breathing difficulties etc) and sensory function.

MMN is a similar condition to CIDP. It is an autoimmune demyelinating neuropathy that leads to slowly progressive asymmetrical weakness that worsens over years without treatment.

IVIg is a recognised treatment for CIDP and MMN. A standard starting dose of 2 g/kg/course, spread over 2-5 days, has been widely used in both research and clinical practice. Due to the chronic nature of CIDP and MMN, most patients with these conditions require repeated doses to avoid relapse, but the frequency of courses and the total dose of IVIg per course required to achieve a steady state varies between patients. Given the modest risks involved with IVIg and its cost, the lowest possible dose and frequency of administration are preferred. Current strategies to reduce dose and frequency involve assessing clinical response to lower doses, but this is both time consuming and imprecise.

DETAILED DESCRIPTION:
The study is designed to slot into normal clinical care, with some extra blood tests performed at times patients would already be attending hospital. An extra blood test is desired 1 week following initial IVIg treatment which would require an extra visit, but this is an optional part of the study.

1. Identification of suitable participant: patient with CIDP or MMN for whom treatment with IVIg has been decided upon by their treating neurologist.
2. Provision of information leaflet and taking of consent. Blood test for Immunoglobulins (Igs), FBC, U&E, LFT and ESR will be taken before initial treatment with 2 g/kg IVIg; this is all part of usual care.
3. 5-30 min following final infusion of first course of IVIg, a blood test for Igs, FBC, U&E, LFT and ESR will be taken.
4. If the patient is willing to make an extra visit 7 days after day 1 of IVIg treatment, they will attend for further Igs, FBC, U&E, LFT and ESR.
5. When the patient attends at 2 weeks for post-IVIg assessment as part of usual care, a blood test for Igs, FBC, U&E, LFT and ESR will be measured again.
6. Usual process of IVIg treatment optimisation will then occur (as practised at the Walton Centre). This is part of usual care, with determination of IVIg dosing interval following clinical optimisation by dose suspension, followed by restabilisation and subsequent dose reductions to determine minimum effective dose.
7. At the 3rd consecutive infusion of IVIg at the minimum effective dose, a pre-IVIg (trough) level of Igs will be taken for the minimum effective IgG level alongside FBC, U&E, LFT and ESR.
8. Statistical analysis looking for correlations between the initial ∆IgG values and the final dose and dosing interval of IVIg will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with CIDP or MMN who are starting Intravenous immunoglobulin in the Walton Centre
* Informed consent

Exclusion Criteria:

* Previous Intravenous immunoglobulin use in the last year

  * Age under 18
  * Lack of mental capacity to consent to treatment or to study participation
  * Concurrent treatment with steroids or other immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with CIDP or MMN starting IVIg under the care of neurologists in The Walton Centre.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Link between IgG levels in the blood of patients with CIDP and MMN | 2 years
  Our primary research objective is to look for a link between ∆IgG levels in the blood of patients with CIDP and MMN following initial IVIg treatment and the ultimate dose required based on clinical response.
  Other blood tests performed at the time of the IgG level include FBC, U&E, LFT and ESR (a measure of plasma viscosity) and will allow a look at the effect of IVIg on these parameters. This could provide clarity as there is much variation in practice as to how often routine blood tests such as FBC, U&E and LFT should be performed in IVIg patients, due to concerns that in some patients there may be biochemical side effects of IVIg treatment. Plasma viscosity may give an indication of risk of thrombotic side effects with IVIg and lead to guidance about, for example, when it is safe to fly after IVIg treatment. Clinical response to treatment will also be recorded
Relationship between IgG and other variables | 2 years
  Secondary analyses of the data collected will look at relationships between ∆IgG and other variables recorded in the data collection. This would include the demographics of the study population, and the severity and type of their disease.

CONTACTS AND LOCATIONS:
Overall Officials: James Holt, Principal Investigator — Walton Centre NHS Foundation Trust
Locations (1):
- The Walton Centre NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No